CLINICAL TRIAL: NCT04614389
Title: Utility of Contrast-Enhanced Sonography and Shear Wave Elastography in Conjunction With ACR TI-RADS for the Evaluation of Thyroid Nodules
Brief Title: Utility of Contrast-Enhanced Sonography and Shear Wave Elastography
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The research team (PI and Sponsor) have agreed that this study would not be feasible to continue.
Sponsor: University of Southern California (Other)
Collaborators: Siemens Medical Solutions USA - CSG (Industry)
Responsible Party: Principal Investigator, Edward Grant, Professor, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HS-19-00296
Record Dates: First submitted 2019-09-25; First posted 2020-11-04 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Thyroid Nodule
MeSH Terms: conditions — Thyroid Nodule

STUDY DESIGN:
Intervention Model Description: Eligible subjects who consent for this study will undergo a SWE and CEUS evaluation of their thyroid gland at the time of their standard of care scheduled thyroid biopsy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- CEUS and SWE (Other): CEUS & SWE
  Interventions: Other: Contrast-enhanced ultrasound; Other: Shear Wave Elastography; Device: Sequoia System

INTERVENTIONS:
Other: Contrast-enhanced ultrasound — Non Invasive Imaging Technique. CEUS involves the use of microbubble contrast agents and specialized imaging techniques to enhance the signal from blood, thus showing flow in macroscopic vessels as well as tissue perfusion informatio
Other: Shear Wave Elastography — Non Ivasive Imaging Technique. Shear Wave Elastography (SWE) is a recently developed technique that uses ultrasound to noninvasively assess the mechanical stiffness of tissue by measuring tissue distortion in ponse to an acoustic radiation force impulse from a focused ultrasound beam.
Device: Sequoia System — UltraSound System Cleared by FDA 510 (k) K180067

SUMMARY:
Our overall hypothesis is that Contrast-enhanced ultrasound (CEUS) and Shear Wave Elastography (SWE) will allow for high diagnostic accuracy of benign and malignant thyroid nodules, which will correlate with and complement the ACR TI-RADS classification system, allowing for more accurate diagnosis of benign and malignant thyroid nodules.

DETAILED DESCRIPTION:
Thyroid nodules are an exceedingly common clinical entity, however, only a small percentage of nodules are malignant. Conventional ultrasound is the current standard for the initial evaluation of thyroid nodules, yet due to several overlapping characteristics between benign and malignant nodules its utility in diagnosis has been limited, leading to a high rate of negative biopsies. To overcome these challenges the American College of Radiology has proposed a Thyroid Imaging Reporting and Data System (TI-RADS) in an effort to decrease unnecessary biopsies [5]. While these efforts have shown encouraging results, further work is still needed. Contrast-enhanced ultrasound (CEUS) and Shear Wave Elastography (SWE) are two emerging non-invasive imaging techniques which have shown promising results in the evaluation of thyroid nodules. However, data is limited and how these imaging modalities could potentially compliment ACR TI-RADS is unknown.

ELIGIBILITY:
Inclusion Criteria:

* - Patients over the age of 18 with one or more thyroid nodules diagnosed on conventional ultrasound within the last 6 months.
* Patients referred for standard of care thyroid nodule biopsy, ordered at the discretion of the treating physician and/or radiologists.
* Patients must demonstrate ability to understand and express willingness to sign a written informed consent to undergo SWE and CEUS imaging prior to their thyroid nodule biopsy.

Exclusion Criteria:

* Patients who are pregnant, nursing, or less than 18 years of age
* Thyroid nodules ≤1 cm

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2021-07-07 (Actual); Study Completion 2021-07-07 (Actual)

PRIMARY OUTCOMES:
Agreement: 1) between two radiologists for visually assessed CEUS result and 2) between the radiologists reconciled visual assessment result and the gold standard result (biopsy). | 8 months
  Kappa analysis will be used to assess the agreement between the two radiologists visual assessment result. The rating result of each radiologist will be compared to the pathological result using Kappa analysis as well.

SECONDARY OUTCOMES:
Agreement between the statistical model predicted result using quantitative metrics from CEUS and/or SWE and the gold standard result (biopsy). | 12 months
  Kappa analysis will be used to re-assess the agreement between the two radiologists visual assessment result. Any disagreement between the radiologists will need to be reconciled and consensus reached. The final assessment result from the radiologists will be compared to the cytology and/or surgical gold standard using anther Kappa test.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Grant, MD, Principal Investigator — University of Southern California
Locations (1):
- USC Department of Radiology, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No